CLINICAL TRIAL: NCT07093749
Title: PATSy Perspectives on Antibiotics and Tracking Symptoms in Children - a Mixed Methods Feasibility Study
Brief Title: Perspectives on Antibiotics and Tracking Symptoms in Children
Acronym: PATSy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 116407
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Urinary Tract Infection; Cellulitis; Impetigo; Pharyngitis; Tonsillitis; Respiratory Tract Infections; Otitis Media
Keywords: Paediatrics; Antibiotics; Digital Health; Infection
MeSH Terms: conditions — Urinary Tract Infections; Cellulitis; Impetigo; Pharyngitis; Tonsillitis; Respiratory Tract Infections; Otitis Media; Infections

STUDY DESIGN:
Intervention Model Description: This is a largely observational study with a small device feasibility portion. The primary outcome of the study is looking at feasibility and satisfaction of study instruments. In addition, approximately 60 of the anticipated total of 300 participants will be invited to wear a Garmin Smartwatch to collect data about heart rate, heart rate variability, skin temperature and sleep and activity levels. Data collected with the Garmin Smartwatch will be compared to parent reported symptoms (collected via surveys) in order to determine level of agreement and investigate if further research into the devices use may be useful.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): All participants eligible participants parent/guardian will be asked to complete:
  1. Daily symptom tracking questionnaires for the duration of their antibiotic course
  2. One-time questionnaire (at enrolment) about parents/guardians' perspectives on antibiotic course duration and stopping antibiotics early
  3. Two short follow up questionnaires (day 14 and day 28) to record if antibiotics have been restarted and for perspectives/concerns and feedback on study instruments and procedures.
  In addition, a small number of participants will also be asked to wear a Garmin Smartwatch for the duration of their antibiotic course (3 devices only available, will be offered when available - approximately 60 participants).
  Interventions: Device: Garmin Smartwatch

INTERVENTIONS:
Device: Garmin Smartwatch — Garmin Venu 3 - Worn for the duration of antibiotic course

SUMMARY:
The study will assess families' perspectives and decision-making regarding the duration of oral antibiotic courses prescribed to children (4-17 years) who present with uncomplicated bacterial infections at the Royal Children's Hospital (RCH) Emergency Department (ED). The study will involve (i) children discharged from ED on oral antibiotics and (ii) children transferred to Hospital-in-the-Home (HITH) on IV antibiotics who then switch to oral antibiotics. In addition, the study will assess how feasible and acceptable it is to track children's symptoms via the Garmin Smartwatch and the WeGuide platform (WeGuide is a patient engagement software platform that allows for enrolment, consent, and data collection [via questionnaires/surveys and from the Garmin Smartwatches] through a singular platform).

DETAILED DESCRIPTION:
This is a mainly observational study looking at the feasibility and acceptability of the study instruments and procedures to be incorporated into an upcoming clinical trial. Parents/guardians will be asked to provide feedback on study procedures and questionnaires. The study will also assess feasibility and acceptability of a shorter course of antibiotic therapy (i.e. stopping earlier) to be tested in the upcoming clinical trial (noting that no antibiotics will be stopped early in this study).

The study will also include a clinical trial component. A small number of participants will be invited to wear a Garmin Smartwatch to collect data about heart rate, heart rate variability, skin temperature and sleep and activity levels. Data collected with the Garmin Smartwatch will be compared to parent reported symptoms (collected via the questionnaires noted above) in order to determine the level of agreement.

All study surveys and Garmin data will be collected through the WeGuide platform. WeGuide is a patient engagement software platform that allows for enrolment, consent, and data collection (via questionnaires/surveys and from the Garmin Smartwatches) through a singular platform.

Study participants will be children (4-17 years of age) who present to the RCH with uncomplicated bacterial infections and are prescribed oral antibiotics (either immediately or as switch from IV antibiotics after transfer to HITH) as standard of care, to assess their and their parents' satisfaction with the study instruments employed in this study, in preparation for the upcoming clinical trial.

WeGuide and Garmin are supporting the PATSy study through the WeGuide and Garmin Health Grant for Digital Health and Wellbeing. The grant includes use of the WeGuide platform and the Garmin Trackers. WeGuide and Garmin have no role in recruitment, data collection, data analysis or publication of the study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of ≥ 4 years and ≤ 17 years at enrolment.
* Diagnosed with any of the following at RCH ED: urinary tract infection (UTI), cellulitis, impetigo, pharyngitis, tonsillitis, respiratory tract infections, otitis media.
* Prescribed oral antibiotics (either immediately or as switch from IV antibiotics after transfer to HITH) as standard of care due to having uncomplicated infection as deemed by their treating doctor.
* Parent/guardian provides a signed and dated informed consent form.

Exclusion Criteria:

- Parent/guardian does not speak English

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of days Garmin Tracker was worn during antibiotic course | Baseline through to Day 10
  Participants will wear the Garmin Tracker for the duration of their antibiotic course. Number of days Garmin Tracker worn collected via WeGuide app. WeGuide is a patient engagement software platform that allows for enrolment, consent, and data collection (via questionnaires/surveys and from the Garmin Smartwatches) through a singular platform.
Number of parents/participants who report issues (via study-specific questionnaire) with Garmin Tracker use | Day 10
  As reported in the daily symptom questionnaires completed by parent/guardian via WeGuide.
Number of parents/participants who report issues (via study-specific questionnaire) with Garmin Tracker use | Day 14
  As reported in the day 14 follow-up questionnaire completed by parent/guardian via WeGuide.
Issues with Garmin Tracker use (as recorded on study-specific questionnaires) - reports by frequency | Day 14
  As reported in the day 14 follow-up questionnaire or the daily symptom questionnaires completed by parent/guardian via WeGuide.
Acceptability of the Garmin Tracker as measured by a study-specific targeted questionnaire | Day 14
  As reported in the day 14 follow-up questionnaire completed by parent/guardian via WeGuide.
Percentage of completed study-specific questionnaires | Baseline through to Day 28
  All study specific questionnaires completed by parent/guardian via WeGuide
Number of parents/participants who report issues completing study-specific questionnaires | Day 10
  As reported in the daily symptom questionnaires completed by parent/guardian via WeGuide.
Number of parents/participants who report issues completing study-specific questionnaires | Day 28
  As reported in the follow-up questionnaire completed by parent/guardian via WeGuide.
Issues with completing questionnaires (as recorded on study-specific questionnaires) - reports by frequency | Day 10
  As reported in the daily symptom questionnaires completed by parent/guardian via WeGuide.
Issues with completing questionnaires (as recorded on study-specific questionnaires) - reports by frequency | Day 28
  As reported in the follow-up questionnaires completed by parent/guardian via WeGuide.
Number of parents/participants who expressed no concerns with study procedures | Day 28
  As reported in questionnaires completed by parent/guardian via WeGuide.
Acceptability of the study procedures as measured by a study-specific targeted questionnaire | Day 28
  Targeted questions will be asked to the parent/guardian to elicit feedback on study experience. Open-ended questions analysed via thematic analysis, closed-ended questions assessed as a percentage of each response.
Number of parents willing to be contacted regarding joining a parent group | Day 28
  Parents will be asked if they are willing to be contacted regarding participation in an upcoming parent group. The parent group will helps us understand parent/child points of view in antibiotic research and provide consumer input into the development of the upcoming clinical trial.
Number of parents/participants who completed all study-specific procedures | Day 28
  All study-specific procedures completed by parent/guardian via WeGuide - includes questionnaires and Garmin Tracker use (for those participants that are invited to and consent to wearing)

SECONDARY OUTCOMES:
Agreement between reports of fever recorded by the Garmin Tracker versus the daily questionnaire - measured using Cohen's kappa coefficient | Baseline to Day 10
  As assessed by Garmin Tracker and study-specific daily questionnaires completed by parent/guardian via WeGuide
Agreement between reports of sleep quality recorded by the Garmin Tracker versus the daily questionnaire - measured using Cohen's kappa coefficient | Baseline to Day 10
  As assessed by Garmin Tracker and in study-specific daily questionnaires completed by parent/guardian via WeGuide
Agreement between reports for activity level recorded by the Garmin Tracker versus reports of daytime lethargy/tiredness in the daily questionnaire | Baseline to Day 10
  As assessed by Garmin Tracker and in study specific daily questionnaires completed by parent/guardian via WeGuide
Number of participants who re-start antibiotics within 28 days of antibiotic commencement as reported in study-specific questionnaire | Day 28
  As reported in the study-specific day 28 follow-up questionnaire completed by parent/guardian via WeGuide.
Number of participants who are still unwell at Day 28 as reported in study-specific questionnaire | Day 28
  As reported in the study-specific day 28 follow-up questionnaire completed by parent/guardian via WeGuide.
Number of participants who finished complete course of antibiotics as reported in study-specific questionnaire | Day 14
  As reported in the study-specific day 14 follow-up questionnaire completed by parent/guardian via WeGuide. Participant who finished complete course of antibiotics is defined as a participant whose parent reports that all prescribed doses are administered exactly as prescribed in the study specific questionnaire delivered via WeGuide
Number of reported doses of antibiotics administered versus doses prescribed as reported in study-specific questionnaire | Day 10
  As reported in study-specific daily questionnaires completed by parent/guardian via WeGuide
Number of participants who report stopping antibiotics early due to resolution of symptoms - as reported on the study-specific questionnaire | Day 14
  Stopping antibiotics early as reported in day 14 follow-up questionnaire completed by parent/guardian via WeGuide. Symptom resolution defined as normalisation of Garmin Tracker health parameters or parent/guardian reporting of no symptoms in daily symptom questionnaire completed via WeGuide.
Reason for stopping antibiotics early as reported on study-specific questionnaire | Day 14
  As reported in the study-specific day 14 follow-up questionnaire completed by parent/guardian via WeGuide.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results that are published after de-identification (text, tables, figures and appendices) will be made available long-term for use by future researchers from a recognised research institution who meet access criteria as outlined below.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months following analysis and publication of the subsequent planned clinical trial.
Access Criteria: Researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre